CLINICAL TRIAL: NCT06290583
Title: Comparison Between the Effect of Spinal Bupivacaine Versus Spinal Prilocaine on Maternal Blood Pressure in Cesarean Section
Brief Title: Comparing the Effect of Spinal Bupivacaine Versus Spinal Prilocaine on Maternal Blood Pressure in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gaber Ahmed, Lecturer in anesthesiology, intensive care and pain management, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Prilocaine in cesarean section
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Spinal Anesthetics Causing Adverse Effects in Therapeutic Use
MeSH Terms: interventions — Bupivacaine; Prilocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group B (Active Comparator): Patients will be given spinal anesthesia with bupivacaine (10 mg) added to morphine (100 microgram) and will be diluted with 0.9% saline to the 3 ml final volume to be injected.
  Interventions: Drug: Bupivacaine
- Group P (Active Comparator): Patients will be given spinal anesthesia with prilocaine (50 mg) added to morphine (100 microgram) and will be diluted with 0.9% saline to the 3 ml final volume to be injected.
  Interventions: Drug: Prilocaine

INTERVENTIONS:
Drug: Bupivacaine — Spinal anesthesia with standard dose of bupivacaine
  Other Names: Intrathecal Bupivacaine
  Arms: Group B
Drug: Prilocaine — Spinal anesthesia with 50 mg dose of Prilocaine.
  Other Names: Intrathecal prilocaine
  Arms: Group P

SUMMARY:
one of the most common complications associated with spinal anesthesia is hypotension, which can have adverse effects on both the mother and the fetus. The present study compare prilocaine versus bupivacaine in spinal anesthesia on hypotension and there effect on maternal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant >36 weeks singleton baby
* American Society of Anesthesiologists (ASA) physical status 2
* Age : between 18 years old and 35 years old

Exclusion Criteria:

* Pregnant women with cardiac disease and history of psychiatric illness
* Pregnant women who received spinal anesthesia and converted to general anesthesia
* Women who have sensitivity to local anesthetics,
* Women who have Eclampsia, abruption placenta or placenta previa
* Women who have coagulopathy, thrombocytopenia with platelet count less than 80,000/cm3, myasthenia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Maternal arterial blood pressure | at base line before induction and every 3 minute during the first 15 min after spinal then every 5 mins until the end of surgery and every 1 hour postoperatively for 6 hours
  Noninvasive blood pressure will be measured at selected time frame.. Hypotension will be defined as a decrease of systolic blood pressure of at least 20% from baseline. Upon its occurrence, and/or appearance of nausea and dizziness, treatment will be immediately with ephedrine 5mg/ dose

SECONDARY OUTCOMES:
Evaluation of duration of motor block | will be assessed before skin incision and every 15 min intervals until the end of surgery and then at 30-min intervals until its complete regression
  the time to motor block regression (duration of motor block), defined as the time between complete block (score 1) after induction of prilocaine or bupivacaine and no motor block (score 6) on the Modified Bromage scale (1, complete motor block; 2, almost complete motor block, ability to move the feet only; 3, ability to move the knees; 4, ability to raise the leg but unable to keep it raised; 5, ability to keep the leg raised for 10 s; 6, no weakness).
Total dose of ephedrine | From beginning of administration of spinal anesthesia until complete regression of motor blockade
  When hypotension occurred postspinal ephedrine 5mg per dose will be given to restore blood pressure to 90% of its baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G Ahmed, MD, Principal Investigator — Lecturer in anesthesiology, intensive care and pain management, South Valley University
Locations (1):
- South Valley University, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No